CLINICAL TRIAL: NCT04382261
Title: Impact of Periodontal Bacteria at Baseline on the Effectiveness of Periodontal Therapy Outcomes in Patients With Periodontitis: A Prospective Clinical and Microbial Study
Brief Title: Impact of Periodontal Bacteria at Baseline on the Effectiveness of Periodontal Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Messina (Other)
Responsible Party: Principal Investigator, Gaetano Isola, DDS, PhD, Researcher, University of Messina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-2018-10
Record Dates: First submitted 2020-05-06; First posted 2020-05-11 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periodontitis quadrant (Placebo Comparator): Patients undergo non surgical quadrant scaling and root planing
  Interventions: Procedure: Scaling and root planing
- Periodontitis full mouth (Active Comparator): Patients undergo non surgical full mouth scaling and root planing
  Interventions: Procedure: Scaling and root planing

INTERVENTIONS:
Procedure: Scaling and root planing — Full mouth or quadrant SRP

SUMMARY:
In light of the controversy that are already approved but that however still exists regarding the efficacy and influence of the protocols for the management of Periodontitis, the aim of this study was to evaluate, at 6 months follow-up, the post-treatment clinical parameters and immunological and gingival microbial profiles in patients with periodontitis, treated by either SRP in addition to full mouth scaling or quadrant scaling

DETAILED DESCRIPTION:
This trial was conducted in accordance with the World Medical Association's Declaration of Helsinki of 1975, and reviewed in 2008. The local ethical committee of the University of Messina approved the study protocol and each patient was carefully informed about the possible inherent risks of the study and provided their informed written consent 102 patients, , aged 27 to 65 (mean age 44.2) were assessed for eligibility. In all subjects, subgingival plaque was acquired from 4 separate proximal sites at 180 days after therapy.

ELIGIBILITY:
Inclusion Criteria:

1. good condition of general health,
2. a minimum of 2 teeth for each quadrant with a Pocket Depth (PD) ranging from 4-6 mm,
3. no involvement of the furcation,
4. a minimum of a six teeth per quadrant, respectively.

Exclusion Criteria:

1. periodontal therapy during the last 12 months,
2. assumption of antibiotics during the last 6 months,
3. pregnancy,
4. any systemic condition which might affect the effects of the study treatment,
5. previous or current radiation or immunosuppressive therapies,
6. use of mouthwash containing antimicrobials during the previous 3 months,
7. no use of hormonal contraceptives,
8. medication by anti-inflammatory and immunosuppressive drugs,
9. previous history of hard-drinking,
10. smoking,
11. class II and III tooth mobility.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Clinical Attachment level | 180 days
  Analysis of reduction of clinical attachment level

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Isola, Study Chair — University of Messina
Locations (1):
- University of Messina, Messina, Italy

IPD SHARING:
Plan to Share IPD: Yes
Sharing inflammatory results
Supporting Information: Study Protocol
Time Frame: 1 year
Access Criteria: University website and pubmed